### NCT03519204

**Study ID:** VOLBELLA-005

**Title:** A randomized, multicenter, no-treatment-controlled study of the safety and effectiveness of JUVÉDERM® VOLBELLA® with Lidocaine for lip enhancement in Chinese adults

Statistical Analysis Plan Date: 16-July-2018

### 1. Title Page

#### STATISTICAL ANALYSIS PLAN

A randomized, multicenter, no-treatment-controlled study of the safety and effectiveness of JUVÉDERM® VOLBELLA® with Lidocaine for lip enhancement in Chinese adults

Study Number: VOLBELLA-005

Development Phase: Pivotal

Product Name: JUVÉDERM® VOLBELLA® with Lidocaine injectable

gel

Sponsor: Allergan Information Consulting (Shanghai) Co., Ltd.

**Suite 5605** 

56F, 1266 West Nanjing Road

Jingan District

Shanghai, China, 200040

This document is the property of Allergan, Inc. and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan, Inc.

# 2. Table of Contents

| 1. | Title | Page | | | 1 |
|---|---|---|---|---|---|
| 2. | Tabl | e of Co | ntents | | 2 |
| | 2.1 | List o | f Tables | | 3 |
| 3. | | | | and Definition of Terms | |
| 4. | intro | | | | |
| | 4.1 | Study | | ummary | |
| | | 4.1.1 | Overall | Design | 7 |
| | | 4.1.2 | | r of Subjects | |
| | 4.2 | Study | Objective | es and Endpoints | 8 |
| 5. | Stati | stical N | <b>lethodolo</b> | gy and Study Endpoints | 14 |
| | 5.1 | Statist | cical and A | Analytical Plans | 14 |
| | | 5.1.1 | | on Conventions | |
| | | | 5.1.1.1 | Analysis Populations | |
| | | | 5.1.1.2 | Study Treatments | |
| | | | 5.1.1.3 | Statistical Methodology | |
| | | | 5.1.1.4 | Missing Data | |
| | | | 5.1.1.5 | Site Pooling | |
| | | 5.1.2 | Demogr | raphics | 16 |
| | | | 5.1.2.1 | Analysis Populations | 16 |
| | | | 5.1.2.2 | Subject Disposition | 16 |
| | | | 5.1.2.3 | Protocol Deviations | 17 |
| | | | 5.1.2.4 | Demographics | 17 |
| | | | 5.1.2.5 | Baseline Characteristics | 17 |
| | | | 5.1.2.6 | Medical History | 18 |
| | | | 5.1.2.7 | Prior and Concomitant Medications | 18 |
| | | | 5.1.2.8 | Exposure to Study Treatment | 18 |
| | | | 5.1.2.9 | Administration of Study Treatment | 19 |
| | | 5.1.3 | Effectiv | reness Analyses | 19 |
| | | | 5.1.3.1 | Primary Effectiveness Endpoint | |
| | | | 5.1.3.2 | Secondary Effectiveness Endpoints | 20 |
| | | 5.1.4 | • | Analyses | |
| | | | 5.1.4.1 | Study Treatment Exposure and Compliance | 22 |

Table 5-2

Table 5-3

| | | | 5.1.4.2 | Adverse Events | 22 |
|---|---|---|---|---|---|
| | | | 5.1.4.3 | Injection Site Responses (ISR) | 23 |
| | | | 5.1.4.4 | Procedural Pain | 24 |
| | | | 5.1.4.5 | Clinical Laboratory Assessments | 24 |
| | | | 5.1.4.6 | Vital Signs and Physical Measurement | 24 |
| | | | 5.1.4.7 | Electrocardiograms | 24 |
| | | | 5.1.4.8 | Pregnancy Test Analyses | 25 |
| | | 5.1.5 | Subgrou | up Analyses | 25 |
| | | 5.1.6 | Interim | Analyses | 25 |
| | 5.2 | Deter | mination | of Sample Size | 25 |
| | 5.3 | Chang | ges in the | Conduct of the Study or Planned Analyses | 25 |
| | | 5.3.1 | Change | s in the Conduct of the Study | 25 |
| | | 5.3.2 | Change | s to Analyses Prior to Database Lock | 26 |
| 6. | Data | Handli | ing and A | nalysis Conventions | 26 |
| | 6.1 | Analy | sis Days | | 26 |
| | | 6.1.1 | Missing | g/Incomplete Treatment End Date | 27 |
| | 6.2 | Analy | | Windows | |
| | | 6.2.1 | Effectiv | /eness | 27 |
| | | 6.2.2 | | | |
| | 6.3 | Missi | ng/Incom | plete Date Conventions | 28 |
| | | 6.3.1 | Missing | g/Incomplete AE Start Date | 28 |
| | | 6.3.2 | Missing | g/Incomplete AE End Date | 29 |
| | 6.4 | Imput | ted Value | Listing Conventions | 29 |
| 2.1 | l | L | ist of Ta | ables | |
| Tal | ole 3-1 | A | Abbreviati | ons and Definitions of Terms | 6 |
| Tol | ala 4-1 | C | tudy Obje | eatives and Corresponding Endnaints | 0 |
| Tal | ole 4-1 | <u></u> | iuuy Obje | ectives and Corresponding Endpoints | 0 |
| Tal | ole 5-1 | A | analysis P | opulations | 14 |

| Table 5-4 | Analysis Population | 16 |
|---|---|---|
| Table 5-5 | Subject Disposition Summaries | 17 |
| Table 5-6 | Protocol Deviation Summary | 17 |
| Table 5-7 | Demographic Summaries | 17 |
| Table 5-8 | Baseline Characteristics Summaries | 17 |
| Table 5-9 | Medical History | 18 |
| Table 5-10 | Medication | 18 |
| Table 5-11 | Exposure to Study Treatment | 19 |
| Table 5-12 | Administration of Study Treatment | 19 |
| Table 5-13 | Effectiveness Assessments | 20 |
| Table 5-14 | Effectiveness Endpoint Baseline Definitions | 20 |
| Table 5-15 | Primary Effectiveness Analyses | 20 |
| Table 5-16 | Secondary Effectiveness Analyses | 21 |
| Table 5-18 | AE Terms | 22 |
| Table 5-19 | AE Summaries | 23 |
| Table 5-20 | ISR Analyses | 23 |
| Table 5-21 | Procedural Pain Analyses | 24 |
| Table 5-22 | Physical Examination Analyses | 24 |
| Table 5-23 | Subgroup Analyses. | 25 |
| Table 5-24 | Sample Size Assumptions | 25 |
| Table 6-1 | Analysis Day Definitions | 26 |
| Table 6-2 | Effectiveness Analysis Visit Definitions for Treatment Group | 27 |
| Table 6-3 | Effectiveness Analysis Visit Definitions for Control Group during Control | ol Period |

| Table 6-3 | Effectiveness Analysis Visit Definitions for Control Group during Treatment | |
|---|---|---|
| | Period | 28 |

# 3. List of Abbreviations and Definition of Terms

Table 3-1 Abbreviations and Definitions of Terms

| Abbreviation/Term | Definition |
|-------------------|-------------------------------------------------|
| 3D | 3-dimensional |
| AE | Adverse event |
| ATC | Anatomical therapeutic chemical |
| CFB | Change from baseline |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| eCRF | Electronic case report form |
| EI | Evaluating Investigator |
| EKG | Electrocardiogram, electrocardiographic |
| ISR | Injection Site Response |
| ITT | Intent-to-treat |
| LFS | Lip Fullness Scale |
| LOCF | Last observation carried forward |
| MedDRA | Medication Dictionary for Regulatory Activities |
| mITT | Modified intent-to-treat |
| PP | Per-protocol |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| TI | Treating Investigator |
| TP | Treated period |
| UCP | Untreated control period |
| WHO | World health organization |

#### 4. Introduction

This statistical analysis plan (SAP) details comprehensive, technical specifications of the statistical analyses of the effectiveness and safety data outlined and/or specified in the final protocol of Study VOLBELLA-005 (Amendment 2 dated 2015-07-29). This SAP will be approved prior to database lock.

### 4.1 Study Design Summary

# 4.1.1 Overall Design

This is a randomized, multicenter, no-treatment-controlled study of the safety and effectiveness of JUVÉDERM® VOLBELLA® with Lidocaine for lip enhancement in Chinese adults. Subjects will be randomized at a 3:1 ratio either to have treatment with VOLBELLA with Lidocaine at the outset of the study (VOLBELLA with Lidocaine group, also referred to as the treatment group, or VOLBELLA group) or to have treatment delayed by 3 months (no-treatment control group, also referred to as the control group). Subjects with Lip Fullness Scale (LFS) score of Minimal, Mild, or Moderate as assessed by Evaluating Investigator (EI) will be enrolled in the study based on inclusion criteria. Randomization will be stratified by baseline LFS score (ie, LFS score rated as Minimal, Mild, or Moderate at the randomization visit by EI).

Treatment and safety assessments of a subject throughout the study will be performed by the same Treating Investigator(TI) (maximum 2 TIs per site), and effectiveness assessments will be performed by the same EI. The EI will remain blinded to treatment assignments throughout the duration of the study.

For subjects randomized to the treatment group, the study treatment will be on the same day as randomization (or within 30 days after screening). Subjects may undergo an optional touch-up treatment at the day 30 visit after initial treatment, if the TI assesses that optimal correction was not achieved. Routine follow-up visits for safety and effectiveness will occur at 1, 3, and 6 months after the last treatment (initial or touch-up treatment, whichever is last). Long-term safety data will be collected by telephone call at 9 and 12 months after the last treatment.

Meanwhile, subjects randomized to the no-treatment control group will attend study visits at months 1 and 3 of the no-treatment control period. After the completion of the control period, control group will receive optional treatment and optional touch-up treatment. Routine follow-up visits will occur at 1, 3, and 6 months. Safety follow-up phone call will be at 9 months.

At initial treatment visit, the TI will inject the treatment into the vermilion body, vermilion border (including the Cupid's bow), and philtral columns, as needed for lip enhancement. The

subject will rate procedural pain on an 11-point scale immediately after receiving the injections, and the TI will assess the ease of injection and the product moldability. Subjects will complete a safety diary for 30 days and will receive a safety follow-up telephone call at 3 days after each initial and touch-up treatment.

## 4.1.2 Number of Subjects

Up to 176 subjects will be randomized at up to 9 Chinese sites.

### 4.2 Study Objectives and Endpoints

The objective of this study is to evaluate the safety and effectiveness of VOLBELLA with Lidocaine for lip enhancement in a Chinese population.

Each study primary objective and secondary objective are presented with corresponding endpoint(s) below:

Table 4-1 Study Objectives and Corresponding Endpoints

| Objectives | Endpoints |
|---|---|
| To evaluate and compare the effectiveness of<br>Volbella with no-treatment control in lip<br>enhancement among Chinese population | <ul> <li>Primary Endpoint</li> <li>Responder at Month 3 (Subject showing ≥ 1-point improvement (increase in fullness)) in LFS score compared with baseline as assessed by EI</li> </ul> |
| | <ul> <li>Secondary Endpoint(s)</li> <li>Responder at Month 3 (Subject showing ≥ 1-point improvement (increase in fullness)) in LFS score compared with baseline as assessed by subject</li> <li>Change from baseline to month 3 in overall lip volume as measured from 3D images</li> <li>Percentage change from baseline to month 3 in lip surface area as measured from 3D images</li> </ul> |
| To evaluate the safety of Volbella in lip<br>enhancement among Chinese population | Safety Assessments • Study treatment exposure • Adverse events (AE) • Injection site responses (ISR) • Procedural pain • Clinical laboratory values (routine hematology and blood chemistry testing and urinalysis) |

| <ul> <li>Vital sign</li> <li>Physical measurement</li> <li>EKG</li> <li>Urine pregnancy test</li> </ul> |
|---|
|---|









# 5. Statistical Methodology and Study Endpoints

# 5.1 Statistical and Analytical Plans

Subjects will receive treatment at the outset of the study (treatment group) or have treatment delayed by 3 months (control group). The analysis based on period up to Month 3 is referred to as "Untreated Control Period" (UCP). After the control group receives treatment, safety and effectiveness data will be collected. The analysis period based on treatment group and control group after treatment will be referred to as "Treated Period" (TP).

Statistical analyses will be conducted using SAS Version 9.3 or newer.

#### **5.1.1** Common Conventions

#### **5.1.1.1 Analysis Populations**

The analysis populations will consist of subjects as defined below:

Table 5-1 Analysis Populations

| Population | Definition | Study Treatment |
|---|---|---|
| Modified Intent-to-<br>Treat (mITT)<br>population | <ul> <li>All subjects who are randomized to study treatment (treatment group) and receive at least 1 study device treatment and have baseline and at least 1 post-treatment assessment of the primary variable</li> <li>All subjects who are randomized to the no-treatment control group and have baseline and at least 1 follow-up assessment of the primary variable</li> </ul> | As treated |
| Per-protocol (PP)<br>population | All mITT subjects who have baseline LFS score of Minimal, Mild, or Moderate, have Month 3 LFS assessments, and do not have any significant protocol deviations affecting the primary effectiveness endpoint | As treated |
| Safety population | <ul> <li>All subjects randomized to the treatment (treatment group) who receive at least 1 study treatment</li> <li>All subjects randomized to the control group</li> </ul> | As treated |

Subjects will be analyzed as treated. All effectiveness analyses will be performed using the mITT population. Additional sensitivity analyses for the primary effectiveness analysis will also be performed using PP population. All safety analyses will be performed using the safety population.

# **5.1.1.2 Study Treatments**

The following treatment groups are defined for this study:

- Study treatment: VOLBELLA with Lidocaine injectable gel
- Control Treatment: No-treatment control

# 5.1.1.3 Statistical Methodology

The methodologies defined below apply as specified to individual endpoints defined in this SAP.

Table 5-2 Statistical Methodology

| Methodology | Description |
|---|---|
| Categorical counts | Number of subjects in individual categories |
| | <ul> <li>Subjects with ≥ 1 qualifying event counted once per individual category</li> </ul> |
| | <ul> <li>N included = subjects with non-missing value for by-visit analysis</li> </ul> |
| Categorical | <ul> <li>Number and percentage of subjects in individual categories</li> </ul> |
| descriptives | <ul> <li>Subjects with ≥ 1qualifying event counted once per individual category</li> </ul> |
| | <ul> <li>N included = subjects with non-missing value for by-visit analysis</li> </ul> |
| Event descriptives | <ul> <li>Number and percentage of events in individual categories</li> </ul> |
| | <ul> <li>Events counted individually for each instance</li> </ul> |
| | <ul> <li>Percentage denominator = total number of events</li> </ul> |
| Continuous | • N included, mean, standard deviation (SD), Q1, median, Q3, minimum, maximum |
| descriptives | <ul> <li>N included = subjects with non-missing value</li> </ul> |
| CFB descriptives | <ul> <li>Continuous descriptives for baseline, postbaseline, and change from baseline<br/>(CFB) values</li> </ul> |
| | <ul> <li>N included = subjects with non-missing values at both baseline and the specified<br/>postbaseline analysis visit</li> </ul> |
| CFB 2-sample t-test | Continuous descriptives for baseline, postbaseline, and CFB values |
| • | For comparing VOLBELLA group vs. no-treatment control group during UCP |
| | (Volbella minus control) |
| | <ul> <li>Mean differences</li> </ul> |
| | <ul> <li>P-values and 95% CI from 2-sample t-test</li> </ul> |
| | <ul> <li>N included = subjects with non-missing values at both baseline and the specified</li> </ul> |
| | postbaseline analysis visit |
| CFB Wilcoxon test | <ul> <li>Continuous descriptives for baseline, postbaseline, and CFB values</li> </ul> |
| | <ul> <li>For comparing VOLBELLA group vs. no-treatment control group during UCP</li> </ul> |
| | (Volbella minus control) |
| | o Mean differences |
| | P-values and 95% CI from Wilcoxon rank-sum test |
| | <ul> <li>N included = subjects with non-missing values at both baseline and the specified<br/>postbaseline analysis visit</li> </ul> |
| Responder exact test | <ul> <li>Categorical descriptives for responders</li> </ul> |
| | <ul> <li>Exact binomial 95% CI of percentages within group</li> </ul> |
| | <ul> <li>For comparing VOLBELLA group vs. no-treatment control group during UCP</li> </ul> |
| | (VOLBELLA minus control) |
| | <ul> <li>Responder rate difference</li> </ul> |
| | <ul> <li>95% exact unconditional confidence interval</li> </ul> |
| | <ul> <li>P-value from 2-sided Fisher's exact test</li> </ul> |
| | <ul> <li>N included = with non-missing values at both baseline and the specified<br/>postbaseline analysis visit</li> </ul> |
| Responder exact | Categorical descriptives for responders |
| 95% CI within | Exact binomial 95% CI of percentages within group |
| group (treatment | N included = with non-missing values at both baseline and the specified |
| group only) | postbaseline analysis visit |
| Responder CMH | Categorical descriptives for responders |

| Methodology | Description |
|---|---|
| test | Responder rate differences for VOLBELLA group vs. no-treatment group during UCP |
| | <ul> <li>P-values from Cochran-Mantel-Haenszel test stratified by baseline characteristic comparing VOLBELLA group vs. no-treatment group during UCP</li> <li>N included = with non-missing values at both baseline and the specified postbaseline analysis visit</li> </ul> |

# 5.1.1.4 Missing Data

General missing data handling conventions are summarized as follows:

Table 5-3 Missing Data Handling by Endpoint Type

| <b>Endpoint type</b> | Timing | Missing Data Handling |
|---|---|---|
| Responder | Month 3 UCP | All subjects included (mITT population) |
| | | <ul> <li>Multiple imputation with 5 imputed datasets is applied to</li> </ul> |
| | | subjects with Month 3 LFS missing using the below model: |
| | | Month 3 LFS = $\beta_0 + \beta_1$ Baseline LFS + $\beta_2$ Month 1 LFS |
| Responder | Month 3 UCP | All subject included (mITT population) |
| | | <ul> <li>Last observation carried forward (LOCF) for subjects with</li> </ul> |
| | | Month 3 LFS missing, baseline value will be carried forw |
| | | if no postbaseline value before Month 3 |
| | | Last observation will be carried forward regardless of schedule/ |
| | | unscheduled visit or analysis window flag. |

The above missing data handling conventions will only be used for sensitivity analysis of the primary effectiveness endpoint.

# 5.1.1.5 Site Pooling

No site pooling will be done. All analyses will also be presented by investigational site. No inferential statistics will be presented for by site analyses.

# **5.1.2 Demographics**

# **5.1.2.1** Analysis Populations

The distribution of subjects within the analysis populations will be summarized as follows:

Table 5-4 Analysis Population

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| All Screened | List of all screened | Screening and | Listing |
| | | Baseline screening | |
| mITT, PP and Safety | Distribution in total and by treatment | After randomization | Categorical counts |
| populations | group | | |

## 5.1.2.2 Subject Disposition

Subject disposition encompasses the distribution of subjects who enter, complete, and discontinue during each specified analysis period, along with eCRF-reported discontinuation reasons from each respective analysis period. Subject disposition will be summarized as follows:

Table 5-5 Subject Disposition Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Study disposition | Distribution in the randomized subjects in | Month 3, final | Categorical |
| | total and by treatment group | | descriptives |

#### **5.1.2.3** Protocol Deviations

Protocol deviations will be defined in a separate document, including significance classification. Protocol deviations will be presented as follows:

Table 5-6 Protocol Deviation Summary

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Significant protocol | Number (%) of subjects with significant | During study period | Categorical counts |
| deviations | protocol deviations | | |

### 5.1.2.4 Demographics

Demographics will be summarized for mITT population in total and by treatment group as follows:

Table 5-7 Demographic Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Age | Age (years) relative to informed consent date | Informed consent | Continuous descriptives |
| Sex | <ul> <li>Race <ul> <li>Male</li> <li>Female</li> </ul> </li> <li>Race <ul> <li>Asian</li> </ul> </li> <li>Ethnicity</li> <li>Chinese</li> </ul> | Screening | Categorical counts |

#### **5.1.2.5** Baseline Characteristics

Baseline characteristics will be summarized in total and by treatment group for the mITT populations as follows:

Table 5-8 Baseline Characteristics Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| LFS score as assessed | Number (%) of subjects in each category | Screening | Categorical |
| by EI | (Minimal, Mild, Moderate, Marked, Very | _ | descriptives |
| | Marked) | | |

| LFS score as assessed by Subject | Number (%) of subjects in each category (Minimal, Mild, Moderate, Marked, Very Marked) | Randomization | Categorical descriptives |
|---|---|---|---|
| Fitzpatrick skin phototype | Number (%) of subjects in each category (I, II, III, IV, V, VI, as well as I/II, III/IV, V/VI) | Screening | Categorical descriptives |
| Exposure to Sunlight (hrs per day) | Exposure to Sunlight (hrs per day) | Screening | Continuous descriptives |
| Smoking status | Number (%) of subjects in each category, current, former, and never smoke | Screening | Categorical counts |
| Duration of smoking (in years) | Duration of smoking (in years) | Screening | Continuous descriptives |

### **5.1.2.6 Medical History**

Medical history, encompassing abnormalities and surgeries reported as occurring before the Screening Visit, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 18.1 or newer. Unique subjects who report medical history events will be presented as subject listing for the Safety Population.

Table 5-9 Medical History

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Abnormalities and | Abnormalities and surgeries occurring | Screening | Listing |
| surgeries | before the Screening Visit | | |

#### **5.1.2.7** Prior and Concomitant Medications

Medications will be coded using the World Health Organization (WHO) Drug Dictionary, version March 2014 or newer. Unique subjects who reported medications (Anatomical Therapeutic Chemical (ATC) 4 class and PT) will be presented as subject listing for the Safety Population.

Table 5-10 Medication

| Endpoint | | Description | Timing | Methodology |
|---|---|---|---|---|
| Treatment | Prior medications | Medications taken before the study treatment | Screening | Listing |
| Group | | regardless of medication end date | | |
| | Concomitant | Medications taken on or after the study treatment and | UCP | Listing |
| | medications during | before Safety Day 91 (at month 3), regardless of | | |
| | UCP | medication start date or end date | | |
| | | (For treatment group, concomitant medications during | | |
| | | UCP consist a subset of concomitant medications | | |
| | | during TP.) | | |
| | Concomitant | Medications taken on or after the study treatment | TP | Listing |
| | medications during TP | regardless of medication start date | | |
| Control | Prior medications | Medications taken before randomization regardless of | Screening | Listing |
| Group | | medication end date | | |
| | Concomitant | Medications taken after randomization and before | UCP | Listing |

| Endpoint | | Description | Timing | Methodology |
|---|---|---|---|---|
| | medications | optional treatment (at month 3), regardless of | | |
| | during UCP | medication start date or end date | | |
| | Concomitant | Medications taken on or after the study treatment | TP | Listing |
| | medications during TP | regardless of medication start date | | |

## **5.1.2.8** Exposure to Study Treatment

Treatment exposure related variable will be summarized for safety population by treatment group (treatment group and treated control group), treatment (combined initial and touch-up, initial, touch-up), and treatment area as in Table 5-11. For treated control group, data after receiving initial treatment at Month 3 are included.

Table 5-11 Exposure to Study Treatment

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Volume injected | Summarize by treatment group, | Initial, | Continuous |
| • Total | treatment, and treatment area | Touch-up | descriptives |
| Upper Lip | | | |
| <ul> <li>Lower Lip</li> </ul> | | | |
| Philtral Columns | | | |
| Treatment sites | Summarize by treatment group, | Initial, | Categorical counts |
| • Total | treatment, and treatment area | Touch-up | |
| Upper Lip | | | |
| <ul> <li>Vermilion body</li> </ul> | | | |
| <ul> <li>Vermilion border</li> </ul> | | | |
| <ul> <li>Lower Lip</li> </ul> | | | |
| <ul> <li>Vermilion body</li> </ul> | | | |
| <ul> <li>Vermilion border</li> </ul> | | | |
| <ul> <li>Philtral Columns</li> </ul> | | | |

# **5.1.2.9** Administration of Study Treatment

Variables related to administration of treatment will be summarized for safety population by treatment group (treatment group and treated control group), treatment (initial, touch-up), and treatment area as in Table 5-12. For treated control group, data after receiving initial treatment at Month 3 are included.

 Table 5-12
 Administration of Study Treatment

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Pretreatment Anesthesia | Ice, Topical, Injectable, Other | Initial, | Categorical |
| <ul> <li>Pretreatment Anesthesia type</li> </ul> | | Touch-up | counts |
| Pretreatment Anesthesia duration (minutes) | Anesthesia duration is computed as | Initial, | Continuous |
| <ul> <li>Pretreatment Anesthesia duration</li> </ul> | injection time minus start of anesthesia | Touch-up | descriptives |
| | administration time. | | |
| | Summarize by treatment group, | | |
| | treatment, and anesthesia type. | | |
| Treatment administration | Summarize by treatment group, | Initial, | Categorical |
| <ul> <li>Injection technique</li> </ul> | treatment (initial or touch-up), and | Touch-up | counts |
| <ul> <li>Planes of injection</li> </ul> | treatment area | | |
| <ul> <li>Needle gauge length</li> </ul> | | | |

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Pretreatment Anesthesia | Ice, Topical, Injectable, Other | Initial, | Categorical |
| <ul> <li>Pretreatment Anesthesia type</li> </ul> | | Touch-up | counts |
| Pretreatment Anesthesia duration (minutes) | Anesthesia duration is computed as | Initial, | Continuous |
| Pretreatment Anesthesia duration | injection time minus start of anesthesia administration time. | Touch-up | descriptives |
| | Summarize by treatment group, | | |
| | treatment, and anesthesia type. | | |
| Massage used | | | |
| <ul> <li>Device/Needle problem or</li> </ul> | | | |
| malfunction | | | |
| Characteristics of the product | Summarize by treatment group, | Initial, | Categorical |
| <ul> <li>Injection ease</li> </ul> | treatment (initial or touch-up), and | Touch-up | counts |
| <ul> <li>Product moldability</li> </ul> | treatment area | | |

# **5.1.3** Effectiveness Analyses

All effectiveness analyses will be based on the mITT Population.

The following effectiveness assessments are defined as:

Table 5-13 Effectiveness Assessments

| Assessment | Description |
|---|---|
| Lip fullness | Assessed by EI and subject based on the overall lip fullness using the 5-point LFS. |
| | (Vey Marked, Marked, Moderate, Mild, Minimal) |
| Overall lip volume | The volume of the overall lips as measured from 3D images. |
| Lip surface area | The lip surface area as measured from 3D images. |

Baseline assessments for applicable effectiveness endpoints are defined as follows:

**Table 5-14 Effectiveness Endpoint Baseline Definitions** 

| Endpoint | Description | Timing |
|---|---|---|
| Overall Lip fullness | Baseline refers to the last evaluation prior to initial treatment | Screening/ |
| <ul> <li>Overall lip volume</li> </ul> | for treatment group, and prior to randomization for control | Randomization |
| <ul> <li>Lip surface area</li> </ul> | group | |
| <ul> <li>Philtral column</li> </ul> | | |
| definition | | |

# **5.1.3.1** Primary Effectiveness Endpoint

The primary effectiveness analysis based on UCP is summarized in the following table. Subjects with baseline LFS score as assessed by EI of Minimal, Mild, or Moderate are enrolled in the study. A LFS (as accessed by EI) responder is defined as a subject with at least one grade improvement from baseline on 5-point LFS as assessed by EI.

Table 5-15 Primary Effectiveness Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| LFS Responder as | Superiority of VOLBELLA with | Month 3 | Responder exact |
| assessed by EI | Lidocaine over no-treatment control | | test |
| | Number (%) of responders by treatment group (mITT population) | | |

The primary effectiveness analysis will be performed based on the mITT population without any missing data imputation. For treatment subjects, assessments within window will be used. For control subjects who do not receive optional treatment, the assessments within month 3 window will be used. For control subjects who receive optional treatment, the assessments within month 3 window and before optional treatment will be used. Sensitivity analysis will be performed using missing data handling conventions as described in Section 5.1.1.4 as well as using PP population.

### **5.1.3.2** Secondary Effectiveness Endpoints

The secondary effectiveness analysis based on UCP is summarized in the following table.

Table 5-16 Secondary Effectiveness Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| LFS responder as | Number (%) of responders by treatment | Month 3 | Responder exact |
| assessed by subject | group | | test within group |
| | | | (treatment group |
| | | | only) |
| Change from baseline in | Summary by treatment group | Month 3 | CFB 2-sample t- |
| overall lip volume | | | test or Wilcoxon |
| | | | test |
| Percentage change from | Summary by treatment group | Month 3 | CFB 2-sample t- |
| baseline in lip surface | | | test or Wilcoxon |
| area | | | test |







# 5.1.4 Safety Analyses

Safety analyses will be based on the Safety Population.

# **5.1.4.1** Study Treatment Exposure and Compliance

See Sections 5.1.2.8 and 5.1.2.9

#### 5.1.4.2 Adverse Events

The following treatment emergent adverse event (TEAE) terms are defined:

Table 5-18 AE Terms

| Term | Description | Timing |
|---|---|---|
| Treatment | An event that initially occurs or increases in severity on or after the treatment and before | UCP |
| group | safety day 91 (month 3) | |
| | (For treatment group, TEAEs during UCP consist a subset of TEAEs during TP.) | |
| | An event that initially occurs or increases in severity on or after the treatment | TP |
| Control | An event that initially occurs or increases in severity on or after randomization and | UCP |
| Group | before optional treatment at month 3 | |
| | An event that initially occurs or increases in severity on or after optional treatment at | TP |
| | month 3 | |

AEs, encompassing abnormalities reported as occurring after the Screening Visit, will be coded using MedDRA version 18.1 or newer. A listing for all AEs in the treatment and control groups will be presented. Additionally, unique subjects reporting AEs as well as number of events in the following AE categories will be summarized for treatment subjects, control subjects after treatment, and all treated subjects as listed in Table 5-19. AEs during UCP will be listed only.

Table 5-19 AE Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Overall summary | Treatment-emergent AEs (TEAEs) | TP | Categorical counts, |
| | <ul> <li>Treatment-related TEAEs</li> </ul> | | Event descriptives |
| | <ul> <li>At injection site</li> </ul> | | |
| | <ul> <li>Not at injection site</li> </ul> | | |
| | <ul> <li>All Serious AEs (SAEs)</li> </ul> | | |
| | <ul> <li>Treatment-related SAE</li> </ul> | | |
| | <ul> <li>At injection site</li> </ul> | | |
| | <ul> <li>Not at injection site</li> </ul> | | |
| | <ul> <li>Discontinued due to TEAE</li> </ul> | | |
| | <ul> <li>Deaths</li> </ul> | | |
| TEAEs | <ul> <li>Overall summary and by SOC, PT, and</li> </ul> | TP | Categorical counts, |
| | severity | | Event descriptives |
| Treatment-related | Overall summary and by SOC, PT, and | TP | Categorical counts, |

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| TEAEs | severity | | Event descriptives |
| | <ul> <li>Overall summary by duration, time to</li> </ul> | | |
| | onset, outcome, and treatment required | | |
| SAEs | Overall summary and by PT | TP | Listing |
| AEs leading to | Overall summary and by PT | TP | Listing |
| discontinuation | | | |

Note: SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the treatment group. AEs for control group after optional treatment are summarized.

Time to onset for TEAEs will be computed as

AE start date - reference date + 1,

where the reference date is initial treatment date for TEAEs occurring on or after initial treatment but before touch-up treatment, and the reference date is touch-up treatment date for TEAEs occurring on or after touch-up treatment.

Duration for TEAEs will be computed as AE end date – AE start date + 1.

### 5.1.4.3 Injection Site Responses (ISR)

ISRs recorded in subject diaries after each treatment (initial, touch-up) will be summarized for that treatment by predefined symptoms.

Table 5-20 ISR Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| ISR severity | Maximum reported severity | Initial, Touch-up | Categorical counts |
| ISR duration | Duration from first instance of the symptom to the last instance of the symptom within the treatment period, where last instance means no further symptoms till the end of the 30-day diary period. Duration is derived as date of last ISR minus date of first ISR plus one. | Initial, Touch-up | Categorical counts |
| ISR | All ISR Diary analysis day will be derived using diary date minus last treatment date plus one. | Initial, Touch-up | Listing |

#### 5.1.4.4 Procedural Pain

Subject assessment of procedural pain (pain during injection) on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) after initial treatment will be summarized.

Table 5-21 Procedural Pain Analyses

| | Endpoint | Description | Timing | Methodology |
|---|------------|-------------|--------|-------------|
| - | Liiupoiiit | Description | 1 ming | Michiganogy |

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Procedural pain | Summary of pain scores as continuous | Initial | Continuous |
| | scale | | descriptive |

## **5.1.4.5** Clinical Laboratory Assessments

Clinical laboratory assessments are taken at Screening, Month 1 and Month 6. Subjects with at least one abnormal finding will be listed for the Safety Population.

## 5.1.4.6 Vital Signs and Physical Measurement

Vital signs and physical measurement (height and weight) will be listed and summarized for the Safety Population.

Table 5-22 Physical Examination Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Vital signs | Summary of blood pressure (systolic and diastolic in a sitting position), temperature, pulse, and respiratory rates | Month 1, 3 (UCP),<br>Month 1, 3, 6 (TP) | Continuous descriptives |
| Physical measurement | Summary of height, weight, and BMI | Screening | Continuous descriptives |

#### 5.1.4.7 Electrocardiograms

Electrocardiograms (EKG) will be taken at Screening and initial treatment visit. Subjects with abnormal finding will be listed.

# **5.1.4.8** Pregnancy Test Analyses

Urine pregnancy test is taken at screening, initial, touch-up, and Month 6. Subjects with positive result will be presented as listing.

# 5.1.5 Subgroup Analyses

Subgroup analyses of the primary effectiveness endpoint will be performed by baseline lip LFS score and volume injected ( $\leq$  median vs > median). All analyses will be repeated for each investigational site descriptively.

Table 5-23 Subgroup Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| LFS Responder as | Number (%) of responders by | Month 3 | Categorical count |
| assessed by EI by | treatment group by baseline LFS | | |
| baseline LFS score | score | | |
| LFS Responder as | Number (%) of responders by | Month 3 | Categorical count |

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| assessed by EI by volume | treatment group by volume | | |
| injected | injected (< median, and > | | |
| | median) | | |
| All analyses by | Summary by investigational site | As described in Table | As described in Table |
| investigational site | | 5-15, 5-16, 5-17 | 5-15, 5-16, 5-17 |

## 5.1.6 Interim Analyses

Not applicable.

# **5.2** Determination of Sample Size

Up to 176 subjects will be randomized at up to 9 Chinese sites.

 Table 5-24
 Sample Size Assumptions

| Parameter | Assumption / Estimate |
|---|---|
| Primary endpoint | Lip fullness assessment responder |
| Risk difference <sup>1</sup> | 34.1% (79% Volbella vs 44.1% Control) |
| SD | NA |
| α | 5% |
| Sides | 2 |
| Power | > 96% |
| N per group | 111 in treatment group, 37 in no-treatment control group |
| Drop-out Rate | 15% |
| N total randomized | 176 |

<sup>&</sup>lt;sup>1</sup> Based on interim data from Study JULIDO-002.

## 5.3 Changes in the Conduct of the Study or Planned Analyses

# **5.3.1** Changes in the Conduct of the Study

Prior to database lock, there were no changes in study conduct.

# **5.3.2** Changes to Analyses Prior to Database Lock

Cross table for overall lip fullness responders between subjects and Evaluating Investigators will not be provided.

# 6. Data Handling and Analysis Conventions

# 6.1 Analysis Days

Analysis day for effectiveness, ISR, and AE are defined as follows:

Table 6-1 Analysis Day Definitions

| Term | Description |
|---|---|
| Analysis day: | VOLBELLA Group |
| Effectiveness Day | Relative to the last treatment date (either the initial treatment, if no touch-up is performed, |

| Term | Description |
|---|---|
| | or the touch-up treatment) |
| | If analysis date >= last treatment date: |
| | • Effectiveness Day = analysis date – last treatment date + 1 |
| | • Effectiveness Day 1 = last treatment date |
| | If analysis date < last treatment date: |
| | • Effectiveness Day = analysis date – last treatment date |
| | • Effectiveness Day -1 = day before last treatment date |
| | Control group before receiving treatment |
| | Relative to the randomization date |
| | If analysis date >= randomization date: |
| | • Effectiveness Day = analysis date –randomization date +1 |
| | • Effectiveness Day 1 = randomization date If analysis date < randomization date: |
| | • Effectiveness Day = analysis date –randomization date |
| | Effectiveness Day -1 = day before randomization date |
| | Control group after receiving treatment |
| | Relative to the last treatment date (either the initial treatment, if no touch-up is performed, |
| | or the touch-up treatment) |
| | If analysis date >= last treatment date: |
| | • Effectiveness Day = analysis date – last treatment date + 1 |
| Amalancia dan | Effectiveness Day 1 = last treatment date VOLDELLA Crown |
| Analysis day<br>Safety Day | VOLBELLA Group Relative to the immediate prior treatment data (initial or toyek up) |
| | Relative to the immediate prior treatment date (initial or touch-up) If analysis date >= initial treatment date: |
| | <ul> <li>Safety Day = analysis date – immediate prior treatment date + 1</li> </ul> |
| | <ul> <li>Safety Day 1 = immediate prior treatment date</li> </ul> |
| | If analysis date < initial treatment date: |
| | • Safety Day = analysis date – immediate prior treatment date |
| | • Safety Day -1 = day before immediate prior treatment date |
| | Control group before receiving treatment |
| | Relative to the randomization date |
| | If analysis date >= randomization date: |
| | • Safety Day = analysis date –randomization date +1 |
| | • Safety Day 1 = randomization date |
| | If analysis date < randomization date: • Safety Day = analysis date -randomization date |
| | <ul> <li>Safety Day -1 = day before randomization date</li> </ul> |
| | Treated Control after receiving treatment |
| | Relative to the immediate prior treatment date (initial or touch-up) |
| | If analysis date >= initial treatment date: |
| | • Safety Day = analysis date – immediate prior treatment date + 1 |
| | <ul> <li>Safety Day 1 = immediate prior treatment date</li> </ul> |

# **6.1.1 Missing/Incomplete Treatment End Date**

Not applicable.

# 6.2 Analysis Visit Windows

#### **6.2.1** Effectiveness

The analysis visit windows for effectiveness endpoints are defined as follows:

Table 6-2 Effectiveness Analysis Visit Definitions for Treatment Group

| Analysis Visit | Target Day of the Visit | Analysis Visit Window |
|---|---|---|
| Screening <sup>a</sup> | N/A | Screening visit |
| Baseline | N/A | Randomization/Initial treatment visit |
| Touch-up treatment b | Day 30 After Initial Treatment | Day 30 after initial treatment visit |
| Last treatment c | Day 1 | Day 1 |
| Month 1 | Day 31 | Days [2, 61] |
| Month 3 | Day 91 | Days [62, 136] |
| Month 6 | Day 181 | >=Day 137 |

<sup>&</sup>lt;sup>a</sup> Subjects may have screening and randomization on the same day. In such cases, only randomization visit is relevant.

Table 6-3 Effectiveness Analysis Visit Definitions for Control Group during Control Period

| Analysis Visit | Target Day of the Visit | Analysis Visit Window |
|---|---|---|
| Screening <sup>a</sup> | N/A | Screening visit |
| Baseline | Day 1 | Randomization visit |
| Month 1 | Day 31 | Days [2, 61] |
| Month 3 | Day 91 | From Day 62 to study exit day if the subject didn't receive optional treatment, or to the day of optional treatment if the subject received optional treatment The assessments before the optional treatment on that day will be accounted for Month 3 visit. |

Table 6-4 Effectiveness Analysis Visit Definitions for Control Group during Treatment Period

| Analysis Visit | Target Day of the Visit | Analysis Visit Window |
|---|---|---|
| Baseline | N/A | Randomization visit |
| Initial treatment <sup>a</sup> | N/A | N/A |
| Touch-up treatment <sup>b</sup> | Day 30 After Initial Treatment | Day 30 after initial treatment visit |
| Last treatment <sup>c</sup> | Day 1 | Day 1 |
| Month 1 | Day 31 | Days [2, 61] |

<sup>&</sup>lt;sup>b</sup> Not all subjects will receive touch-up treatment.

<sup>&</sup>lt;sup>c</sup> Initial treatment if touch-up is not performed, otherwise touch-up treatment

| Month 3 | Day 91 | Days [62, 136] |
|---------|---------|----------------|
| Month 6 | Day 181 | >=Day 137 |

<sup>&</sup>lt;sup>a</sup> Initial treatment is at Month 3 visit.

If there are multiple visits occurring within a single visit window with relevant data, the visit closest to the target day listed above will be used in the analysis of the corresponding visit windows regardless of scheduled or unscheduled visit. If two visits are equal distant to the target day and are the same type of visit, then the later visit will be used.

### **6.2.2 Safety**

No analysis visit windows are required for TEAEs and ISRs.

## 6.3 Missing/Incomplete Date Conventions

#### 6.3.1 Missing/Incomplete AE Start Date

Imputation of dates with missing day and/or month is only applied to TEAEs. If adequate information is available, no imputation is needed. TEAE start dates with missing day or month will be imputed as following:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan or the initial treatment date if they have the same year, whichever is later (because TEAE onset is not expected prior to administration of study treatment)
- If day is missing but the month and year are available, then the imputed day will be the first day of the month or the initial treatment date if they have the same month and year, whichever is later

# 6.3.2 Missing/Incomplete AE End Date

Imputation of dates with missing day and/or month is only applied to TEAEs. If adequate information is available, no imputation is needed. TEAE end dates with missing day or month will be imputed as following:

• If day and month are missing but year is available, then the imputed day and month will be 31 Dec or the study exit date if they have the same year, whichever is earlier

<sup>&</sup>lt;sup>b</sup> Not all subjects will receive touch-up treatment.

<sup>&</sup>lt;sup>c</sup> Initial treatment if touch-up is not performed, otherwise touch-up treatment.

• If day is missing but the month and year are available, then the imputed day will be the last day of the month or the study exit date if they have the same month and year, whichever is earlier

# **6.4** Imputed Value Listing Conventions

In general, listings will present the actual partial or missing values rather than the imputed values that may be used in endpoint derivation. In instances where imputed values will be presented, imputed values will be flagged. Actual rules will be fully defined in the table, figure, and data listing specification document.



# **ALLERGAN**

# Statistical Analysis Plan VOLBELLA-005 China

| Date (DD/MMM/YYYY)/Time (PT) | Signed by: | Justification |
|------------------------------|------------|---------------|